CLINICAL TRIAL: NCT03524872
Title: Implant/Abutment Module Stability: a RCT Comparing Original vs Compatible Connections (Estabilidad Del módulo Implante/Pilar: ECA Comparando Conexiones Originales vs Compatibles).
Brief Title: Implant/Abutment Module Stability of Original vs Compatible Connections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Peñarrocha Oltra, Assistanat Postdoctoral Lecturer (Profesor Ayudante Doctor), University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H1497611651778
Record Dates: First submitted 2018-03-03; First posted 2018-05-15 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Bone Loss, Alveolar; Dental Implant Failure Nos
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Anesthesia, Local; Acetaminophen; Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The devices will have the same shape and will be delivered to the surgeon unlabeled in an identical sterile envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Original CAD/CAM abutment (Active Comparator): Patients will be rehabilitated using Sweden&Martina implants and original (Sweden&Martina) CAD/CAM abutments.
  Interventions: Device: Original CAD/CAM prosthetic abutment; Procedure: Local anesthesia; Drug: Painkillers; Drug: Mouthwashes; Device: Implant placement
- Compatible CAD/CAM abutment (Experimental): Patients will be rehabilitated using Sweden&Martina implants and compatible (New Ancorvis) CAD/CAM abutments.
  Interventions: Device: Compatible CAD/CAM abutment; Procedure: Local anesthesia; Drug: Painkillers; Drug: Mouthwashes; Device: Implant placement

INTERVENTIONS:
Device: Original CAD/CAM prosthetic abutment — Original (Sweden&Martina) CAD/CAM abutments will be screwed to the implants at 32N/cm.
  Arms: Original CAD/CAM abutment
Device: Compatible CAD/CAM abutment — Compatible (New Ancorvis) CAD/CAM abutments will be screwed to the implants at 32N/cm.
  Arms: Compatible CAD/CAM abutment
Procedure: Local anesthesia — Infiltration of 4% articaine with 1:100,000 adrenalin (Inibsa).
Drug: Painkillers — Patients will be prescribed ibuprofen 600 mg three times per day for five days
Drug: Mouthwashes — Patients will be prescribed mouth-rinse with chlorhexidine 0.12% twice daily starting 3 days prior to surgery and for 2 weeks afterward
Device: Implant placement — Dental implants (Sweden & Martina, Padua, Italy) will be placed at crestal level and according to the manufacturer's instructions.

SUMMARY:
Together with materials and type of retention, the stability of the implant abutment connection represents one of the key factor for the success rate of an implant supported restoration. The recent diffusion of high quality and easy to use CAD/CAM systems has contributed to market launch of a number of competing companies that offer the so called "clonical" or "compatible" restorative components. Although they are claimed to be identical, the original abutments are supposed to present maximum accuracy and consequently lower microleakage.

The aim of the present randomized controlled trial will be to analyze the implant abutment junction stability comparing implant-supported crowns restored with original components and compatible non-original abutments.

The hypothesis is that original components will present significantly better stability than non-original abutments.

ELIGIBILITY:
Inclusion Criteria:

* Any healthy patient scheduled for an implant-supported restoration will be considered for inclusion in this study, independently of the implant and prosthetic protocols used.

Exclusion Criteria:

* general medical contraindications to oral surgery (American Society of Anesthesiologist, ASA, class III or IV),
* patients <18 years of age,
* smoking habit (>10 cigarettes/day),
* sites with acute infection or requiring regenerative procedures,
* Full Mouth Plaque Score
* Full Mouth Bleeding Score >25 %,
* pregnant and lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Biological complications | 1 year
  Proportion of cases with peri-implant disease.
Biomechanical complications | 1 year
  Proportion of cases with fracture or loosening of screws

SECONDARY OUTCOMES:
Microbial loads | 1 year
  Quantitative analysis of microbial species will be studied using Illumina protocol for 6S ribosomal RNA
Probing Pocket Depth | 1 year
  Measured from the mucosal margin to the bottom of the probable pocket.
Modified Plaque Index | 1 year
  Presence/absence of plaque at the cervical part of the implant-supported crown scored by running a probe along the implant-supported crown surface.
Bleeding on Probing | 1 year
  Presence/absence of bleeding after probing.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Odontológica de la Universitat de Valencia, Fundación Lluis Alcanyis, Valencia, Spain